CLINICAL TRIAL: NCT01582100
Title: Reletex ™ Band as an Adjunct to Standard Therapy in Patients With GERD, Nausea With or Without Vomiting- A Pilot Study
Brief Title: Reletex for Nausea in GERD Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: study was terminated by investigator due to low enrollment
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Pandolfino, Associate Professor of Medicine, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56024
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-07

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GERD subjects with nausea (Experimental): subjects with GERD and nausea will receive treatment with Reletex
  Interventions: Device: Reletex

INTERVENTIONS:
Device: Reletex — Neuromodulation device worn on the wrist

SUMMARY:
Gastroesophageal reflux disease (GERD) is a highly prevalent condition that is frequently encountered in the health care setting. It affects roughly 40% of Americans monthly and 10% weekly. Of those with GERD, there exists a cohort that experience nausea with or without vomiting that is unresponsive to PPI's and anti-emetics. For these patients, treatment options are limited and these symptoms may substantially alter their quality of life. New and novel therapies emerging include neuromodulation devices that may affect the central pathways leading to these symptoms. Of these, the Reletex band has been tested and proven efficacious in the treatment of nausea and vomiting associated with pregnancy, chemotherapy, and surgery, in addition to standard anti-nausea medications. The investigators propose that through a similar mechanism, this device as an adjunct to PPI's and anti-emetics will reduce GERD-associated the nausea with or without vomiting, and by so doing, improve the quality of lives in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 with clinically diagnosed GERD as evidenced by the GerdQ assessment tool and/or ambulatory pH/ pH- impedance monitoring with a component of nausea with or without vomiting.
* Continued symptoms despite a stable dose of FDA approved daily PPI therapy in addition to or without supportive anti-emetics. We will include patients with twice a day PPI dosing, as this is a standard treatment for PPI non-responders.
* Previous gastric emptying study performed as part of the standard care work-up of nausea and vomiting. Patients will be recruited regardless of the results and this information will only be used as a potential predictor for symptom response.

Exclusion Criteria:

* Currently participating in a concurrent clinical trial or completed another trial within past 8 weeks.
* Prior gastrointestinal surgery of the esophagus and stomach.
* Severe esophagitis (Los Angeles esophagitis Grade C and above), Barrett's metaplasia or eosinophilic esophagitis, achalasia or spastic motor disorder
* Unstable medical illness with ongoing diagnostic work-up and treatment. Patients with well-controlled hypertension, diabetes and a remote history of ischemic heart disease that is deemed stable, as judged by the physician-investigator can be included. Current drug or alcohol abuse or dependency.
* Current neurologic or cognitive illness or impairment which would make the patient an unsuitable candidate for hypnosis. This will be determined by the investigators before randomization using the Mini Mental Status Exam in patients with suspected impairment.
* Severe mental illness, e.g., uncontrolled major depression with suicidal ideation, active psychosis, diagnosis of schizophrenia-spectrum disorder.
* Those with nickel, gold, or other metal allergies.
* Those with other neuromodulators or implanted electrical devices such as cardiac pacemakers, AICD's, neurostimulators or transcutaneous electrical nerve stimulation devices (TENS units).
* Females who are or might become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Pandolfino, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Faculty Foundation, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: two subjects were recruited in clinic. One withdrew after experiencing minor wrist discomfort, the other withdrew after determining the visit schedule undesirable.
Groups:
- GERD Subjects With Nausea: Subjects who present with GERD along with nausea (with or without vomiting)
Period: Overall Study
Arm/Group | GERD Subjects With Nausea
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: two subjects with GERD and nausea
Arm/Group | GERD Subjects With Nausea
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea in Patients With GERD
Description: number of events of nausea with or without vomiting in patients with GERD in 4 weeks
Time Frame: 4 weeks
Groups:
- Single Arm Subjects With GERD/Nausea: This is a single arm study measuring the incidence and severity of nausea with or without vomiting in patients with GERD before and after treatment with Reletex
Arm/Group | Single Arm Subjects With GERD/Nausea
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year, 11 months
Groups:
- Wrist Discomfort: subject did not like the feel of the device on wrist
Arm/Group | Wrist Discomfort
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated due to low enrollment. One subject withdrew due to minor wrist discomfort and the other withdrew after determining the study schedule was undesirable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No